CLINICAL TRIAL: NCT00143429
Title: Effect Of Corneal Versus Conjunctival Delivery On The Corneal Safety, Tolerability, and Antihypertensive Efficacy Of The Xalatan Ophthalmic Delivery Device
Brief Title: Corneal Versus Conjunctival Delivery Using a Delivery Device
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A6111127
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2015-03

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

INTERVENTIONS:
Drug: Xalatan

SUMMARY:
Compare the antihypertensive efficacy of three methods for installing Xalatan

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma or ocular hypertension in 1 or both eyes

Exclusion Criteria:

* History of closed/barely open anterior chamber angle or a history of angle closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
IOP level in the study eye

SECONDARY OUTCOMES:
Change in ocular safety assessments. Ocular and systemic adverse events throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer